CLINICAL TRIAL: NCT06156527
Title: A Randomized Phase II Study of LAZE Rti N ib Alone Versus Lazertinib Plus Beva C Izumab for A Dvanced Non Small Cell Lung Cancer With Epidermal Growth Factor Receptor Activating Mutations and Smoking History
Brief Title: A Randomized Phase II Study of LAZE rtiNib Alone Versus Lazertinib Plus bevaCizumab for NSCLC With EGFR + & Smoker
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Beung-Chul AHN, Dr., National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAZENCA Trial
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Lazertinib
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single arm (Active Comparator): lazertinib single arm
  Interventions: Drug: Lazertinib
- combination arm (Experimental): Lazertinib plus bevacizumab
  Interventions: Drug: Lazertinib; Drug: Bevacizumab Injectable Product

INTERVENTIONS:
Drug: Lazertinib — Lazertinib 240mg, QD, daily
  Other Names: Single arm; combinationarm
Drug: Bevacizumab Injectable Product — Bevacizumab: 15mg/kg IV every 3 weeks
  Other Names: combinationarm
  Arms: combination arm

SUMMARY:
Using gefitinib or Osimertinib, an EGFR tyrosine kinase inhibitor (TKI), in patients with active mutations in epithelial cell growth factor receptors (EGFR), 70% response rate (CR+PR) and 90% disease control rate (CR+PR+SD) compared to the current non-small cell therapy, which is significant in the EFRT treatment. However, resistance causes recurrence in most patients. Therefore, it is necessary to develop a more effective treatment. Recently, in Japan, combined allotinib and bevacizumab therapy as primary therapy in non-small cell lung cancer patients with EGFR mutation improved PFS statistically significantly compared to allotinib monotherapy, suggesting the possibility of a new treatment (Hazard ratio 0.605, 95% CI 0.417-0.877, P=0.016). In addition, subsequent osmutinib and bevacizumab combination therapy showed a significant difference in PFS in the smoker group, although they did not show significant improvement in PFS in the entire patient group. (Hazard ratio 0.605, 95% CI 0.417-0.877, P=0.016). Since EGFR mutated lung cancer is highly frequent in Korea, it is necessary to develop more effective treatments for such patients. Therefore, we propose this clinical trial to find out the efficacy of lasertinib and bevacizumab combination therapy.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate PFS of laseratinib and bevacizumab combination therapy as the primary treatment for advanced lung cancer with EGFR mutation.

For laseratinib monotherapy, the expected median PFS is 15 months. On the other hand, assuming the expected median PFS 27 months of laseratinib and bevacizumab combination therapy, the one-sided test alpha level is 0.05, the power 0.8) dropout rate should be approximately 120 (60 people per group) enrolled in this study.

Patients would be enrolled in this study for 18 months and followed up to at least 24 months from the last patient enrollment date.

This study is a phase 2 clinical trial, and the primary goal is PFS, and based on the log rank test, the laseratinib bevacizumab combination therapy group significantly increases PFS when one side p value <0.05.

Fisher's Fisher exact test or chi-square test will be used in consideration of laboratory data and laboratory test abnormalities or clinical adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed patients with locally progressive or metastatic non-small cell lung cancer (IIIB or IV) who have not been diagnosed as squamous cell carcinoma.
2. Patients with one or more measurable lesions in accordance with the RECIST criteria (Version 1.1), tumor lesions located at the previous irradiation site, are considered measurable if progress has been made in those lesions.
3. Patients with institutionalized EGFR mutation (exon 19 deletion or L858R)
4. Patients with a history of smoking, including those who are currently smoking (defined as those who have smoked more than 100 cigarettes in their lifetime)
5. ECOG PS 0-1 Patient
6. Patients with appropriate hematological functions ANC≥1,500/uL, hemoglobin≥9.0g/dL, platelet≥100,000/uL
7. Patients with adequate liver function Total bilirubin < 1 x UNL, AST (SGOT) and ALT (SGPT) < 2.5 x UNL (If there is an interruption: total bilirubin <3 x UNL, AST (SGOT) and ALT (SGPT) <5 x UNL)
8. a patient with appropriate renal function Cr UN UNL, however, can be registered if the creatinine clearance calculated according to the formula Cocroft and Gault is 50 50 ml/min outside the normal range.

   Proteinuria test <2+ (if 22+ then protein 11g must be in 24-hour urine test)
9. Patients with a history of receiving radiation therapy must meet the following criteria.

   - In the case of direct radiation irradiation to the lung lesion area, it must have elapsed at least 12 weeks from the time of registration.
   * In the case of chronic radiation therapy for intracoracic bone metastasis, it must be at least 12 weeks from the time of registration.
   * 2 weeks or more from the time of registration if radiotherapy has been performed on any non-chest area Must be elapsed.
10. At the time of registration, the date of completion of the previous treatment or procedure must pass the period specified below.

    - Surgery (including exploratory/experimental thoracotomy): 4 weeks

    - Pericardial drainage: 1 week

    - pleural adhesion not attributed to anti-species positive substances (including biological response regulators such as Picibanil): 2 weeks

    - Tissue biopsy to confirm selection criteria (including biopsy using thoracoscope): 1 week
    * Procedures for the treatment of trauma (unregistered patients with untreated wounds): 2 weeks
    * Blood transfusion, hematopoietic growth factor administration: 2 weeks
    * The puncture and aspiration cell test: 1 week
    * Administration of other clinical trial medications: 4 weeks
11. Women in childbearing age should be negative in serum or urine pregnancy tests within 7 days prior to test treatment.
12. Male and childbearing female test subjects with female partners' pregnancy must agree to use the following two high-efficiency test methods for at least 180 days after the last dose of the assigned treatment is administered. Bevacizumab can also damage a woman's reproductive ability. Therefore, women who have entered the bevacizumab combination group should be preceded by discussions on preserving the reproductive ability of women who are likely to become pregnant before treatment - asceticism

    - tubal ligation

    - Hormone contraceptives that do not cause drug interactions (such as Mirena)
    * Medroxyprogesterone injection (Depo-Provera)
    * Copper bands and intrauterine devices
    * a partner's vasectomy
    * Partner's use of condoms
13. Patients who have agreed to the clinical trial-

Exclusion Criteria:

- 1) Patients with other malignant tumors except lung cancer within the past three years (except for properly treated cervical epithelial cancer, basal or squamous cell skin cancer, thyroid cancer, and topical prostate cancer surgically treated for healing purposes).

2) Patients with a history of bleeding above Grade 2 (with blood above Grade 2) 2.5mL within 3 months of registration defined as the above bright red blood.) 3) chemotherapy for advanced lung cancer in the past or other systemic anticancer drugs (single-clone antibodies or Patients with tyrosine kinase inhibitors) (However, pre- and post-operative assisted chemotherapy, which ended 6 months before the time of registration, is allowed.) 4) A patient with evidence of invasion of large blood vessels, such as the pulmonary artery or relative vein of a tumor, in contrast examination.

5) Patients scheduled to undergo hydrophobic surgery (including infantile catheter insertion) within 24 hours of the first injection of bevacizumab 6) Current or recent (within 10 days prior to the initial injection of bevacizumab) aspirin (>325 mg/day) and patients with oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (provided that preventive use of anticoagulants is permitted).) 7) Patients currently in use (or unable to discontinue prior to the initial dose of lazertinib) with a drug or natural aid known as a potent CYP3A4 inducer that cannot be discontinued throughout clinical trials before enrollment 8) Any evidence of ILD, drug-induced ILD, past history of radiation interstitial pneumonia requiring steroid treatment, or clinically active ILD 9) Patients undergoing or likely to administer bisphosphonate medication 10) Uncontrolled patients with brain-spinal metastasis (Patients with epilepsy can be registered if they are stabilized asymptomaticly, and treated patients with epilepsy can be registered if they do not currently require steroid treatment.) 11) Patients with clinically significant ophthalmic abnormalities on the surface of the eye (not recommended to use contact lenses) (with corneal perforations or ulcers, symptoms and signs of acute or exacerbated corneal inflammation such as ocular inflammation, tear secretion, blurred vision, eye pain and bleeding) 12) Patients with a history of coagulopathy with hereditary bleeding constitution or risk of bleeding 13) Patients with uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic >100 mmHg) 14) Patients with clinically significant active cardiovascular disease (within 6 months of registration, patients with cerebrovascular accidents and diseases, myocardial infarction, unstable angina, NYHA ClassIIII congestive heart failure, thrombosis, thromboembolism, and severe cardiac arrhythmia that may interfere with drug administration during clinical trials)

The following heart criteria are not limited to one. :

* Average of corrected QT intervals at rest (QTc intervals corrected by Fredericia formula) >470 msec based on QTc values calculated by ECG equipment by the test institution during screening.
* clinically significant abnormal findings found in the rhythm, conduction, or morphology of the ECG at rest (e.g., complete left block, 3rd degree heart block, 2nd degree heart block)
* All factors that increase the risk of QTc prolongation or arrhythmia, including heart failure, hypokalemia, family history of congenital QT prolongation syndrome, sudden death of causes under the age of 40 in the immediate family, combined drugs known to prolong QT spacing and induce Torsades de Points (TdP).

  15) Patients with non-healing wounds, active digestive ulcers, or fractures 16) Patients with active infections and uncontrolled systemic diseases 17) Patients who have a chemical structure similar to lasertinib and bevacizumab or these substances or who have a history of hypersensitivity to active ingredients or inactive excipients of drugs belonging to the family.

  18) Patients who are hypersensitive to CHO (animal cell line from the uterus of Chinese hamsters) cell products or other recombinant human body or humanized antibodies.

  19) Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | every 9 weeks
  Progression -free survival

SECONDARY OUTCOMES:
ORR | every 9 weeks
  Overall Response Rate
OS | 2 years after randomization
  Overall Survival
AE | every 3 weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Beung-Chul AHN, Study Chair — National Cancer Center
Locations (5):
- South Korea (5):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeunggi-do
  - AJOU university hospital, Suwon, Gyeunggi-do
  - Yonsei University Health System, Severance Hospital, Seoul
  - Gangnam Severance Hospita, Seoul

IPD SHARING:
Plan to Share IPD: No